CLINICAL TRIAL: NCT01588431
Title: A Phase II Study of Induction Docetaxel, Cisplatin, Cetuximab and Bevacizumab (TPE-A) Followed by Concurrent Radiation, Cisplatin, Cetuximab and Bevacizumab (XPE-A) in Patients With Locally Advanced Head and Neck Cancer (CTRC# 11-36)
Brief Title: Bevacizumab/Ph 2 for Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 11-36; HSC20120002H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-02-29; First posted 2012-05-01 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Locally advanced head and neck cancer; Squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Cetuximab; Bevacizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (TPE-A) Followed by Concurrent RT(XPE-A), surgery (Experimental): Docetaxel, Cisplatin, Cetuximab and Bevacizumab (TPE-A) Followed by Concurrent Radiation, Cisplatin, Cetuximab and Bevacizumab (XPE-A), surgery
  Interventions: Drug: Docetaxel, Cisplatin, Cetuximab and Bevacizumab (TPE-A) Followed by Concurrent Radiation, Cisplatin, Cetuximab and Bevacizumab (XPE-A), surgery

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, Cetuximab and Bevacizumab (TPE-A) Followed by Concurrent Radiation, Cisplatin, Cetuximab and Bevacizumab (XPE-A), surgery — Induction therapy consists of 3 cycles of bevacizumab 15mg/kg on day 1, cetuximab weekly days 1,8,15 (loading dose of cetuximab 400mg/m2 on cycle 1, day 1, then 250 mg/m2 on all subsequent administrations), cisplatin 75mg/m2 on day 1, docetaxel 75mg/m2 on day 1, repeated every 21 days. After 3 cycles of induction therapy, patients will receive standard radiation 70-74 Gy/ 200 cGy/ daily, 5 days/ week with concurrent weekly cisplatin 30mg/m2, cetuximab 250mg/m2 and bevacizumab 15mg/kg every 3 weeks x 3. There is optional surgery for non-responders in the primary (stable disease) after TPE-A.

SUMMARY:
Locally advanced squamous cell carcinoma of the head and neck (SCCHN) is treated with various combinations of radiation and chemotherapy. This study aims to evaluate the rate of complete responses with induction therapy (primary endpoint) and progression-free survival, overall survival and objective response rates of docetaxel, cisplatin, cetuximab, and bevacizumab (TPE-A) followed by radiation therapy, cisplatin, cetuximab, and bevacizumab (XPE-A). Also, the investigators plan to investigate a panel of EGFR and angiogenesis biomarkers in pre-and post- treatment tumor biopsies. Finally, the investigators will evaluate the associated treatment toxicities and the quality of life.

DETAILED DESCRIPTION:
Locally advanced squamous cell carcinoma of the head and neck (SCCHN) is treated with various combinations of radiation and chemotherapy. Docetaxel and cisplatin have been combined in Phase II trials in recurrent or metastatic head and neck cancer with very encouraging results. Induction therapy with docetaxel/cisplatin followed by chemoradiotherapy was investigated in a randomized Phase II study in nasopharyngeal cancer and showed superior PFS and OS in comparison with chemoradiation alone. Cetuximab is a chimerized EGFR monoclonal antibody that has produced positive results in Phase III trials in combination with either radiation for locally advanced disease or chemotherapy for metastatic disease. Upregulation of vascular endothelial growth factor (VEGF) has been associated with cetuximab resistance. Bevacizumab, an anti-VEGF antibody is currently being investigated in SCCHN with promising results. The investigators have previously shown that cisplatin, docetaxel and cetuximab (TPE) followed by radiotherapy, cisplatin and cetuximab (XPE) is feasible and highly efficacious in locally advanced SCCHN (Argiris, A. et al.JCO 2011). In this Phase II study the investigators evaluate the addition of bevacizumab to induction therapy with TPE (TPE-A) and to subsequent XPE (XPE-A).

Specific aims:

To evaluate the rate of complete responses with induction therapy (primary endpoint) and progression-free survival, overall survival and objective response rates. Also, the investigators plan to investigate a panel of EGFR and angiogenesis biomarkers in pre- and post- treatment tumor biopsies. Finally, the investigators will evaluate the associated treatment toxicities and the quality of life.

Subject population:

The investigators will enroll patients with previously untreated locally advanced SCCHN (see detailed eligibility criteria).

Treatment plan:

Induction therapy consists of 3 cycles of bevacizumab 15mg/kg on day 1, docetaxel 75mg/m2 on day 1, loading dose of cetuximab 400mg/m2 on cycle 1, day 1, then 250 mg/m2 on all subsequent administrations (Day 8 and 15 of cycle 1 and days 1,8,15 of cycles 2 and 3), cisplatin 75mg/m2 on day 1, docetaxel 75mg/m2 on day 1, repeated every 21 days. After 3 cycles of induction therapy, patients will receive standard radiation 70-74 Gy/ 200 cGy/ daily, 5 days/ week with concurrent weekly cisplatin 30mg/m2, cetuximab 250mg/m2 and bevacizumab 15mg/kg every 3 weeks x 3. There is optional surgery for non-responders in the primary (stable disease) after TPE-A.

Statistical design and sample size:

Phase II, two-stage study with complete response rate after induction therapy as the primary endpoint. The sample size is 33 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AJCC 7th edition stage III-IVB head and neck cancer, all sites, including unknown primary tumors.
* Prior to entry in the study the resectability and alternative treatment options for each patient will be determined by a team composed of an Ear, Nose, and Throat Surgeon, a Radiation Oncologist and a Medical Oncologist. Stage determination, optimal local treatment, and its timing according to this protocol will be determined at this evaluation. The unequivocal demonstration of distant metastasis (M1) confers ineligibility.
* Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas, or WHO types I-III of the nasopharynx.
* Unidimensionally measurable disease is required (RECIST 1.1).
* No prior chemotherapy, biologic/molecular targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* Prior surgical therapy will consist only of incisional or excisional biopsy, and organ sparing procedures such as debulking of airway compromising tumors or neck dissection in a patient with an existing primary tumor. Any non-biopsy procedure must have taken place > 4 weeks but < 3 months of initiating protocol treatment.
* ECOG performance status 0-1.
* Age 18 years or older.
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* All patients should have their tumor tissue tested for HPV (in situ hybridization and/or p16 staining by immunohistochemistry), and results must be known prior to study entry, and will consent to have available archival tumor samples, unstained slides or blocks from previous diagnostic or therapeutic procedures submitted for correlative studies, including assessment of target molecules EGFR, VEGF and related biomarkers. Also, patients must agree to submit blood samples for correlative studies at least at baseline.
* Absolute neutrophil count at or above 1500/µl, Platelet count at or above 100,000/µl
* Creatinine clearance 60 ml/min or higher calculated using the Cockcroft-Gault formula:

Calculated Creatinine Clearance = (140-age) X actual body wt (kg)/ 72 X serum creatinine Multiply this number by 0.85 if the patient is female

* Total bilirubin within normal limits and AST/ALT less than 3 times the upper limit of normal.
* Urine dipstick must be < 0-1+ within 2 weeks (14 days) of randomization. If urine dipstick result is > 1+, a calculation of Urine Protein Creatinine (UPC) ratio is required. Patients must have a UPC ratio < 1.0 to participate in the study.

NOTE: UPC ratio of spot urine is an estimation of the 24-urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1gm. UPC ratio is calculated using one of the following formula:

* [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/DI
* [(urine protein) × 0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

  * Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post diagnosis.
  * Patients may not be receiving any other investigational agents.

Exclusion Criteria:

* History of severe allergic reactions attributed to docetaxel or compounds of similar chemical or biologic composition to docetaxel, or other drugs formulated with polysorbate 80.
* Prior severe infusion reaction to a monoclonal antibody or known hypersensitivity to any component of bevacizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study
* No patients with significant baseline sensory or motor neurologic deficits (> grade I neuropathy) will be treated on this study.
* Because patients with immune deficiency are at increased risk of lethal Infections when treated with marrow-suppressive therapy, HIV-positive patients are excluded from the study. Appropriate studies will be undertaken in patients with HIV and those receiving combination anti- retroviral therapies when indicated.
* Patients with HPV positive tumors (P16+ by immunohistochemistry and/or HPV+ by in situ hybridization) AND smoking history =<10 pack-years
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 12 months prior to Day 1
* No history of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (> or = to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Patients should not be on therapeutic anticoagulation therapy (prophylactic use of warfarin 1mg per day is allowed) and INR should be <1.5 at registration
* The use of anti-platelet agents (e.g. dipyridamole (Persatine), ticlopidine (Ticlid), clopidogrel (Plavix)) is allowed only if patient is not receiving aspirin or NSAID's known to inhibit platelet function.
* Major surgical procedure (including neck dissection), open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Pregnant or breast-feeding women will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Wehbe, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Evaluate the rate of complete responses with induction therapy - Change in baseline regarding treatment/tumor response after 3 cycles of chemotherapy (3months); After 8 weeks of chemo + radiation; 1 year up to 10 years. This outcome will be measured with regards to number of participants via RECIST criteria.
Time Frame: 1year up to 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Level of Angiogenesis Biomarkers
Description: Investigate a panel of Epidermal Growth Factor Receptor (EGFR) and angiogenesis biomarkers in pre- and post- treatment tumor biopsies and evaluate the associated treatment toxicities and the quality of life. After 8 weeks of chemo + radiation; 1 year up to 10 years.
Time Frame: 8 weeks up to 10 years
Population: No subjects completed the study, only one subject progressed to long term treatment, but did not survive to 10 years. Biomarkers on tissues were not performed since there were not enough evaluable samples.
Arm/Group | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to 10 years
Arm/Group | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery (N=3)
Decreased White Blood Cell count (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1) — Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (TPE-A) Followed by Concurrent RT(XPE-A), Surgery (N=3)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutrofever (Blood and lymphatic system disorders) | 3 (3)
Decreased platelet count (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Transaminase imbalance (Metabolism and nutrition disorders) | 1 (1)
Low HbA1c (Endocrine disorders) | 3 (3) — Low glycosylated glucose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT01588431/Prot_SAP_000.pdf